CLINICAL TRIAL: NCT06284200
Title: Presence and Comparison of Sarcopenia in Early Rheumatoid Arthritis and Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, Prof. Dr, Kayseri City Hospital
Other Study IDs: sarcopenia eRA
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia
Keywords: Early Rheumatoid Arthritis; Sarcopenia; Rheumatoid Arthritis; Appendicular Skeletal Muscle Mass Index
MeSH Terms: conditions — Sarcopenia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
introduction: In this study, the presence of sarcopenia in cases with early rheumatoid arthritis and established rheumatoid arthritis will be compared.

Materials and Method: According to the power analysis, 24 patients with early rheumatoid arthritis and 24 patients with established rheumatoid arthritis who meet the 2010 American College of Rheumatology (ACR) / European Alliance of Associations for Rheumatology (EULAR) rheumatoid arthritis (RA) classification criteria will be included in the study.

DETAILED DESCRIPTION:
According to the power analysis, 24 patients with early rheumatoid arthritis and 24 patients with established rheumatoid arthritis who met the 2010 ACR / EULAR RA classification criteria will be included in the study. The presence of sarcopenia will be evaluated according to the European Working Group on Sarcopenia in Older People (EWGSOP-2) criteria by performing hand grip strength, muscle mass measurement with Bioelectrical Impedance Analysis (BIA), and 4-meter general walking speed tests. Demographic data of the patients and anti-nuclear antibody (ANA), rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) levels, Simplified Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI), Disease Activity Score ( DAS)28, functional status (health assessment questionnaire (HAQ)), quality of life (RA quality of life scale (RAQoL)), anxiety and depression (hospital anxiety and depression scale (HADS)) results will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the early RA group:

* To be diagnosed with RA according to the 2010 ACR (American Society for the Study of Rheumatism) / EULAR (European Association for the Study of Rheumatism) RA classification criteria
* Being 18 years or older
* Being followed up with a diagnosis of RA for less than 1 year (early RA)

Inclusion criteria for the RA group:

* To be diagnosed with RA according to the 2010 ACR (American Society for the Study of Rheumatism) / EULAR (European Association for the Study of Rheumatism) RA classification criteria
* Being 18 years or older

Exclusion Criteria:

* Presence of other rheumatic disease
* Presence of malnutrition
* Recent surgical history,
* Stroke history,
* Pregnancy,
* Presence of prosthesis or metal implant,
* Presence of a pacemaker,
* Patients over 140 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the planned single-center study, patients with clinically confirmed RA and early RA diagnosed who applied to Kayseri City Hospital Physical Medicine and Rehabilitation outpatient clinic will be included in the study after their consent is obtained.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-03-23 (Estimated); Study Completion 2024-06-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Muscle Mass | once at the baseline
  Muscle mass evaluations in patients will be made using the Bioelectrical Impedance Analysis (BIA) (Multi Frequency Segmental Body Composition) method. According to the data obtained from the BIA device, appendicular skeletal muscle mass index (ASMI). The ASMI cut-off point recommended by the EuropeanWorkingGroup on Sarcopenia in Older People (EWGSOP2) would be <7.26 kg/m2 for men and <5.5 kg/m2 for women. Patients with low ASMI will be evaluated as having sarcopenia.
Evaluation of Muscle Strength | once at the baseline
  In general, hand grip strength is one of two methods used to measure muscle strength in patients with suspected sarcopenia. Hand grip strength is related to strength in other muscles and can therefore be used as a tool to demonstrate muscle weakness. The hydraulic hand dynamometer will be used in all patients included in this study, and measurements will be recorded in kilogram. Measurements will be made with the patient in a sitting position on a chair, with the elbow close to the body and 90 degrees of flexion, and the wrist in neutral.Patients will be asked to grasp the dynamometer as firmly as possible. Three measurements will be taken for the patients and the average was taken. The recommended cut-off point for the hand grip test will be considered to be <27 kg for men and <16 kg for women.Patients with low hand grip strength will be evaluated as having possible sarcopenia.
Evaluation of Muscle Performance | once at the baseline
  Physical performance will be evaluated with a 4-meter general walking speed test. The patient will be asked to walk a distance of 4 meters at his normal pace, as in his daily life, and the time to walk the distance of 4 meters will be calculated in seconds. 4 meter general walking speed will be calculated in m/sec and speeds below 0.8 m/sec will be considered low walking speed.

SECONDARY OUTCOMES:
Rheumatoid Arthritis Quality of Life Scale | once at the baseline
  The Turkish version of the Rheumatoid Arthritis Quality of Life Scale (RAQoL), prepared for use in the Turkish population, is valid, reliable and practical to use in clinical studies. It is recommended that the scale be used in the individual monitoring of patients with RA and in the evaluation of treatment effectiveness in clinical studies.
Health Assessment Questionnaire (HAQ) | once at the baseline
  The HAQ was developed by Fries et al. in 1980 to evaluate the physical limitations of patients with Rheumatoid Arthritis. It gauges activities of daily living consisting of 20 items in 8 sections. Each item is scored between 0-3 (0: no difficulty at all, 1: some difficulty, 2: great difficulty, 3: cannot do it at all). High score means low functionality. The scale was adapted to Turkish society.
Hospital Anxiety and Depression Scale (HADS) | once at the baseline
  Anxiety and depression will measured by using HADS, which is a 14-item questionnaires with 7 responses each for anxiety and depression with a maximum possible score of 3 for a particular response. A score of up to 7 is considered normal, with scores of 8-10 as borderline abnormal and scores 11-21 as being abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: HAVVA TALAY ÇALIŞ, PROF, Study Director — Health Sciences University, Kayseri Medical Faculty
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kocasinan, Kayseri, Turkey (Türkiye)